CLINICAL TRIAL: NCT00946088
Title: Progesterone for Maintenance Tocolysis: A Randomized Placebo Controlled Trial
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: lower than expected enrollment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Deirdre Judith Lyell, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-03312009-2078; 11625 (Other: Stanford University Med. Center IRB)
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone (Active Comparator): Progesterone 400mg per vagina qhs.
  Interventions: Drug: Progesterone
- Polyethylene glycol&hydrogenated vegetable oil (Placebo Comparator): Polyethylene glycol&hydrogenated vegetable oil per vagina
  Interventions: Drug: Polyethylene glycol&hydrogenated vegetable oil.

INTERVENTIONS:
Drug: Progesterone — Progesterone 400 mg per vagina qhs.
  Arms: Progesterone
Drug: Polyethylene glycol&hydrogenated vegetable oil. — Placebo Comparator: Polyethylene glycol 400 distearate & hydrogenated vegetable oil per vagina qhs.
  Arms: Polyethylene glycol&hydrogenated vegetable oil

SUMMARY:
Preterm delivery is the most common cause of infant morbidity and mortality in the United States. Some women have episodes of preterm labor during their pregnancy which can be temporarily stopped. These women, however, are at high risk for delivering before term. At this time, we do not have sufficient evidence to use any medication to help prevent these women from delivering early. Recently, preliminary studies have shown that progesterone may help prevent some women at high risk for preterm delivery from delivering early. Our study will investigate whether progesterone can help this specific group of women, women with arrested preterm labor, deliver healthy infants at term.

DETAILED DESCRIPTION:
The purpose of this study is to test the efficacy of progesterone in prolonging human pregnancies complicated by arrested preterm labor. Animal labor has not been shown to be equivalent to human labor and would not be an appropriate substitute for this study.

In addition, this medication has been previously used in pregnant women without any evidence of significant harm to the mother or fetus. Women will be approached for enrollment in the study during their hospitalization for preterm labor. If they choose to enroll, they will have weekly MD visits at the obstetrical clinic, daily use of vaginal progesterone that will be self administered, and routine obstetric care at the time of recurrent labor and delivery. The daily progesterone is not a part of routine care for these patients. In addition, we will ask patients to fill out a written questionaire one week after starting the medication to describe any subjective symptoms that may be associated with this medication. Finally, we will assess the peripheral levels of progesterone with a blood draw prior to starting the mediation, one week after starting the medication, and at the time of recurrent pre-term labor or delivery. The first two of these blood draws will be in addition to the standard treatment. The final blood draw will involve collecting an extra sample at a time when the participant would normally have blood drawn as a part of routine care.

ELIGIBILITY:
Inclusion Criteria:1. Pregnant women with arrested preterm labor between 24+0 to 33+6 weeks pregnant.

2. Intact membranes 3. Singleton pregnancy 4. Greater than or equal to 18 years of age 5. Cervical dilation less than or equal to 4cm Exclusion Criteria:1. Any contraindication to on-going pregnancy 2. Placental abruption 3. Placenta previa 4. Lethal fetal anomalies 5. Premature rupture of membranes 6. Multiple gestation 7. Less than 18 years old 8. Known allergy to any component of the study medication or placebo 9. Severe maternal medical illness

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2009-10; Primary Completion 2013-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Judith Lyell, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from November 2010 through February 2011.
Groups:
- Polyethylene Glycol 400 Distearate & Hydrogenated Vegetable oi: Polyethylene glycol 400 distearate & hydrogenated vegetable oil
Period: Overall Study
Arm/Group | Progesterone | Polyethylene Glycol 400 Distearate & Hydrogenated Vegetable oi
Started | 4 | 3
Completed | 4 (At least one dose administered and pre-term birth status known.) | 2 (At least one dose administered and pre-term birth status known.)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Polyethylene Glycol & Hydrogenated Vegetable Oil: Polyethylene glycol 400 distearate & hydrogenated vegetable oil
- Total: Total of all reporting groups
Arm/Group | Progesterone | Polyethylene Glycol & Hydrogenated Vegetable Oil | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 28.5 [24 to 33] | 27.0 [19 to 34] | 27.9 [19 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Delivery Rate Prior to 37 Weeks Gestation
Description: Reduction in delivery rate prior to 37 weeks gestation (preterm birth).
Time Frame: Up to 37 weeks of gestation
Measure: Count of Participants; unit: Participants
Groups:
- Polyethylene Glycol&Hydrogenated Vegetable Oil: Polyethylene glycol 400 distearate & hydrogenated vegetable oil per vagina
Arm/Group | Progesterone | Polyethylene Glycol&Hydrogenated Vegetable Oil
Number analyzed (Participants) | 4 | 2
Participants
  Delivery at <37 weeks of gestation | 2 | 0
  Delivery at >=37 weeks of gestation | 2 | 2

2. Secondary Outcome: Maternal Chorioamnionitis
Time Frame: Up to maternal hospital discharge
Measure: Count of Participants; unit: Participants
Groups:
- Polyethylene Glycol & Hydrogenated Vegetable Oil: Polyethylene glycol 400 distearate & hydrogenated vegetable oil per vagina
Arm/Group | Progesterone | Polyethylene Glycol & Hydrogenated Vegetable Oil
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

3. Secondary Outcome: Maternal Anticipated Adverse Medication Reaction
Time Frame: Up to the maternal discharge from delivery hospitalization
Measure: Count of Participants; unit: Participants
Groups:
- Polyethylene & Hydrogenated Vegetable Oil: Polyethylene glycol 400 distearate & hydrogenated vegetable oil per vagina
Arm/Group | Progesterone | Polyethylene & Hydrogenated Vegetable Oil
Number analyzed (Participants) | 4 | 2
Participants | 1 | 0

4. Secondary Outcome: Birthweight
Description: Newborn birthweight in grams
Time Frame: At the time of newborn birth
Measure: Mean (Full Range); unit: grams
Arm/Group | Progesterone | Polyethylene Glycol & Hydrogenated Vegetable Oil
Number analyzed (Participants) | 4 | 2
grams | 2740 [1390 to 3720] | 3275 [3070 to 3380]

5. Secondary Outcome: Neonatal Intensive Care Unit (NICU) Admission
Time Frame: At time of neonatal discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Progesterone | Polyethylene Glycol & Hydrogenated Vegetable Oil
Number analyzed (Participants) | 4 | 2
Participants | 2 | 0

6. Secondary Outcome: Neonatal Morbidity
Time Frame: Up to 28 days after neonatal birth
Measure: Count of Participants; unit: Participants
Arm/Group | Progesterone | Polyethylene Glycol & Hydrogenated Vegetable Oil
Number analyzed (Participants) | 4 | 2
Participants | 1 | 0

7. Secondary Outcome: Neonatal Mortality
Time Frame: Up to 28 days after neonatal birth
Measure: Count of Participants; unit: Participants
Arm/Group | Progesterone | Polyethylene Glycol & Hydrogenated Vegetable Oil
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

8. Secondary Outcome: Neonatal Congenital Abnormalities
Time Frame: Up to the time of neonatal discharge from the delivery hospital
Measure: Number; unit: Neonates
Arm/Group | Progesterone | Polyethylene Glycol & Hydrogenated Vegetable Oil
Number analyzed (Participants) | 4 | 3
Neonates | 0 | 0

9. Secondary Outcome: Number of Days Delay of Delivery
Description: Number of days from intervention to delivery
Time Frame: Up to the time of delivery
Population: exact delivery data unavailable for one term participant
Measure: Median (Full Range); unit: days
Arm/Group | Progesterone | Polyethylene Glycol & Hydrogenated Vegetable Oil
Number analyzed (Participants) | 4 | 2
days | 38.0 [6 to 62] | 47.5 [43 to 52]

ADVERSE EVENTS:
Time Frame: Up to 28 days after the delivery.
Groups:
- Active Comparator: Progesterone: Progesterone 400mg per vagina qhs.
- Placebo Comparator: Polyethylene Glycol&Hydrogenated Vegetab: Placebo Comparator:Polyethylene glycol&hydrogenated vegetable oil per vagina.
Arm/Group | Active Comparator: Progesterone | Placebo Comparator: Polyethylene Glycol&Hydrogenated Vegetab
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

LIMITATIONS AND CAVEATS:
Very limited enrollment, study terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No